CLINICAL TRIAL: NCT00436787
Title: Pharmacokinetic Properties of Fondaparinux Sodium in Morbidly Obese Volunteers
Brief Title: Investigation Into the Therapeutic Dosage of Fondaparinux Sodium, a Medication Used to Prevent Blood Clots in Morbidly Obese Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ART108029
Expanded Access: Available
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Venous Thrombosis; Pulmonary Embolism
Keywords: Anticoagulation Prophylaxis; Venous Thrombosis; Deep Vein Thrombosis; Pulmonary Embolism; Fondaparinux Sodium; Arixtra; Pharmakinetics
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux Sodium

SUMMARY:
Morbidly obese individuals are at high risk for potentially life threatening blood clots around the time of abdominal surgical procedures. Fondaparinux sodium (Arixtra) is an FDA- approved medication used in the prevention of deep venous thrombosis (DVT) at the time of orthopedic or abdominal surgery, as well as for the treatment of DVT and pulmonary embolism (PE). As with many medications, therapeutic dosages have not been fully investigated for the morbidly obese population. Our goal is to study the therapeutic blood levels, after 2 different dosages of the medication are given to morbidly obese volunteers. We will recruit 21 morbidly obese (Body Mass Index (BMI) > 35) individuals who are in the evaluation process for bariatric surgery. They will be divided into 7 groups: 3 participants with BMI 35 - 39.9, 3 with a BMI of 40 - 49.9, 3 with a BMI of 50 - 59.9, 3 with a BMI > 60, 3 with a weight of 100 - 149 KG, 3 with a weight of 150 - 199 KG and 3 with a weight of 200 - 249 KG. Participants will be administered two different doses of the medication with a 2-week interval in between, then blood will be drawn in various intervals throughout the next 48 hours to see which dose provides the best therapeutic levels. Participants will be monitored closely for any side effects or complications.

DETAILED DESCRIPTION:
Bariatric surgery carries a mortality rate of 0.5-1%, with PE found to be the most frequent postoperative complications and causes of death. Currently employed prophylactic methods include unfractionated or low molecular weight heparins in combination with mechanical calf compression. However, despite the implementation of these standard measures, the reported incidence of fatal PE has ranged from 0.2 to 0.64% accounting for between 30 to 50% of deaths after bariatric surgery.

With a reported 40,000 bariatric surgical procedures in 2001, and the numbers growing rapidly every year, there is clearly a need for a more effective prophylaxis from DVT and PE. The pentasaccharide fondaparinux is an anti-thrombotic agent used in the prophylaxis of venous thromboembolism after orthopedic or abdominal surgery. Its clinical value has been established in multiple randomized double blind studies in high-risk major orthopedic surgery where it showed a 55% greater reduction in DVT episodes compared to enoxaparin (Lovenox®) Although fondaparinux has been administered in obese patients in clinical studies for prevention of venous thromboembolism after orthopedic surgery and preliminary results show no influence of ABW on the clinical outcome, the pharmacokinetic properties of the drug in the morbidly obese have not been investigated. Previously published fondaparinux pharmacokinetic studies excluded patients whose body weight was more than 30% of ideal, with the heaviest group being 77.2+/-10.1 Kg and with a BMI of 25.7+/2.6 Kg/m2. Similar studies on low molecular weight heparins, such as enoxaparin and dalteparin, showed predictable anti-Xa activity with weight-based dosing in the morbidly obese.

There has been no study on the pharmacokinetics of this drug in the morbidly obese (BMI>35 Kg/m2). It is clinically imperative to have a predictable anti-Xa level and a predictable DVT prophylactic effect in the morbidly obese whose body weight may vary by as much as 3 to 4 fold higher compared to the average 70 Kg adult. This has become a critical issue in view of the large number of bariatric surgical operations being undertaken, which has increased 150% in the last two years.

The purpose of this study is to assess the pharmacokinetic properties of fondaparinux in morbidly obese volunteers. This is a prospective crossover, randomized study with a 2-week washout period comparing two dosing regimens of fondaparinux in morbidly obese volunteers.

ELIGIBILITY:
INCLUSION

1. Age 19-65 years
2. BMI 35-65 Kg/m2
3. Pregnancy test Negative on day of study
4. Past DVT/PE/MI These patients will not be excluded providing they are not on current therapy with anticoagulants, aspirin, or anti-platelet agents.

EXCLUSION

1. BP ≥ 160/90
2. Temperature > 37.5 0C (99.5 0F)
3. Nursing mothers Exclude if nursing
4. Pregnancy test Positive on day of study
5. Medications Anticoagulants, anti-platelet agents, aspirin, NSAIDs within a month of the study

Past medical history

1. cerebrovascular accident (including TIA within 6 months of the study)
2. Diabetic retinopathy proven by fundoscopy
3. History of inherited thrombotic/hypercoagulable defect
4. Active peptic ulcer disease diagnosed by upper endoscopy
5. Known bleeding disorder, thrombophilia
6. History of heparin induced thrombocytopenia
7. History of bacterial endocarditis
8. Known hypersensitivity to fondaparinux
9. Ulcerative colitis
10. History of GI bleeding
11. History of hematuria
12. Recent surgery (last 3 months)
13. Recent trauma (last 3 months)

Laboratory values

1. Platelet count ≤ 100,000 mm3
2. Hemoglobin < 12 g/dL (women), or < 14 g/dL (men)
3. Prothrombin time > 13 sec
4. PTT > 35 sec
5. ALT 3xULN and bilirubin 1.5xULN (>35% direct); or ALT 5xULN; or ALT 3xULN if associated with the appearance or worsening of hepatitis symptoms or rash
6. Estimated urinary creatinine clearance ≤ 50 ml/min
7. Hematuria on urine dipstick

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2007-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic properties of fondaparinux sodium in morbidly obese individuals.

SECONDARY OUTCOMES:
Comparisons of the pharmacokinetic parameters of morbidly obese participants receiving 2.5 mg or 5 mg dose of fondaparinux sodium with those of healthy normal-weight volunteers established from previous studies.
Comparison of the pharmacokinetic parameters of the 2.5 mg and 5 mg dosage of fondaparinux sodium.
Evaluate the effect of BMI and ABW on the pharmacokinetic parameters of the 2.5 mg and 5 mg dosages of fondaparinux sodium.
Assess the safety of fondaparinux sodium, as measured by defined safety endpoints, and compare the 2 dose groups for differences in the incidence of adverse events (AE).

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Raftopoulos, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Shadyside Medical Building, Pittsburgh, Pennsylvania